CLINICAL TRIAL: NCT00790283
Title: Assessment of the Numen Stent With Evaluation in a Randomized Study
Acronym: ANSWERS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Biomedical Systems S.p.A. (Industry)
Responsible Party: Nader Shehata, International Biomedical Systems S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBS/04-2007; 2008-A00111-54
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Lesion
Keywords: Treatment of de novo lesions in native coronary arteries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Numen (Experimental)
  Interventions: Device: PTCA with stent implantation
- Vision/MiniVision (Active Comparator)
  Interventions: Device: PTCA with stent implantation

INTERVENTIONS:
Device: PTCA with stent implantation — Eligible patients will be randomly assigned to the implantation of one (or more) Numen or Vision/Mini Vision stent.
  Each patient will undergo a 1-month follow-up and a clinical visit at 6 months from the procedure.

SUMMARY:
The purpose of this study is to Evaluate the Short-Term and Mid-Term Safety and Efficacy of the NUMEN Cobalt-Chromium coronary stent for the treatment of de novo lesions in native coronary arteries and compare it to the VISION/MINIVISION coronary stent

DETAILED DESCRIPTION:
The success of bare metal coronary stenting is limited by the restenosis phenomenon, with rates depending on patient vascular morphology and lesion-related factors, the indication for and technique of stent deployment, and others. Drug-eluting stents (DES) improve the treatment of many coronary artery lesions by significantly reducing in-stent restenosis. However, there have numerous limitations resulting from the need for long-term dual antiplatelet therapy, the consequent bleeding risk (old patients, surgery, colon or gastric cancer, trauma), the unknown side-effects of long-term antiplatelet therapy, the cost associated with a long-term thienopyridine regimen, the body's reaction to the stent polymer, and the 0.2% per year increase in late stent thrombosis in comparison with bare metal stents (BMS).

For these reasons, continuous research is devoted to improve the effectiveness of bare metal stents. The ideal stent should be non-thrombogenic, with a low rate of restenosis and late thrombotic events. The NUMEN stent has been designed to meet these criteria, using an extremely low stent strut thickness.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical or instrumental documentation of stable/unstable myocardial ischemia or angina with a >50% lesion on a major coronary vessel and/or side branch > 2.0 mm
* Lesion length ≤ 20 mm
* Vessel requiring stent size with diameter ≥ 2.5 mm

Exclusion Criteria:

* Age < 18 years
* Life expectancy < 6 months
* Chronic renal failure (serum creatinine > 2 mg %)
* Ongoing acute myocardial infarction
* Left ventricular ejection fraction (LVEF) <30%
* Cardiogenic shock
* Documented or suspected systemic and/or infectious disease
* Hypersensitivity to cobalt chromium or contrast media
* Anti-thrombotic drug intolerance
* Cardiac and/or extracardiac documented disease requiring surgical repair
* Patient is not an acceptable candidate for emergent coronary artery bypass surgery
* Primary or secondary pulmonary hypertension (by echo-doppler)
* Planned > 2 stent implantation (except bail-out)
* Recent (< 6 months) PCI or CABG
* Other type of stent implantation (also in case of bail-out)
* Visible endocoronary thrombosis
* Diffuse, severe coronary calcifications
* Use of debulking devices
* Extreme vessel tortuosity
* Unprotected left main stenosis (ULM)
* Bifurcation lesion
* In stent restenosis (ISR)
* Saphenous vein graft (SVG) and arterial by pass (internal mammary artery,IMA)
* Chronic total occlusion (CTO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of Major Adverse Cardiac Events (MACE), Cerebrovascular Events CVE) and Major Bleedings (according to TIMI classification) | 6 months

SECONDARY OUTCOMES:
Any death, cardiac death, stent related fatal / non fatal MI, TVR | 1 month
Any death, cardiac death, stent related fatal / non fatal MI, TVR | 6 months
Cardiac death, fatal/non fatal MI | In hospital
Procedural success, TLR, TVR, ST | In hospital

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Corcos, MD, FACC, Principal Investigator — Clinique Turin, Paris, France
Locations (8):
- France (8):
  - CHU Cote de Nacre, Caen
  - CMC De Parly II, Le Chesnay
  - Clinique Valmente, Marseille
  - Centre Hospitalier Privé Beauregard, Marseille
  - Clinique Vert Coteau, Marseille
  - Clinique Turin, Paris
  - Clinique Alleray-Labrouste, Paris
  - Clinique Saint Gatien, Tours